CLINICAL TRIAL: NCT06335810
Title: Reducing Obesity Using Social Ties (ROBUST): Randomized Control Trial
Brief Title: Reducing Obesity Using Social Ties Program
Acronym: ROBUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 23-10026599; R01DK135949-01 (NIH)
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Weight Loss; Undermining; Communication
MeSH Terms: conditions — Obesity; Weight Loss; Communication

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social Network Intervention (Experimental): Participants will complete 3 communication skills sessions with their social network members during weeks 3, 5, and 15.
  Interventions: Behavioral: Social Network Intervention
- Individual Lifestyle Intervention (Placebo Comparator): Participants will complete standard diabetes prevention program (DPP) based health coaching sessions during weeks 3, 5, and 15.
  Interventions: Behavioral: Individual Lifestyle Intervention
- Social Network Member (Other): Social Network Members will complete 3 communication skills sessions with the social network intervention participant during weeks 3, 5, and 15.
  Interventions: Other: Social Network Member

INTERVENTIONS:
Behavioral: Social Network Intervention — Social Network interventions are an intentional effort to modify or use the characteristics of social networks to improve, generate, and maintain healthy behaviors among individuals and populations. This study will focus on implementing a behavioral social-network intervention to promote changes in weight loss behaviors.
  Arms: Social Network Intervention
Behavioral: Individual Lifestyle Intervention — The individual lifestyle intervention will serve as the control group and will implement the use of DPP based health coaching sessions to promote individual level changes in weight loss behaviors.
  Arms: Individual Lifestyle Intervention
Other: Social Network Member — The social network member will serve as the friend, family member, or co-worker nominated to participate in the social network intervention by the social network intervention participant.
  Arms: Social Network Member

SUMMARY:
This trial aims to test the feasibility and acceptability of addressing interpersonal barriers to weight-related behavior change. Specifically, the study will test if, by including up to two friends, family members, or co-workers in a lifestyle intervention for weight loss, the person enrolled in the study loses more weight than someone whose friends, family members, or co-workers were not invited to participate.

DETAILED DESCRIPTION:
The investigators will evaluate whether the ROBUST intervention not only addresses individual-level behaviors (i.e., healthy eating, increased physical activity) but also:

1. reduces social undermining as well as changes perceived health norms by activating communal coping - a behavioral process that involves thinking, communicating, and acting as if a health risk (i.e., Type 2 diabetes) is shared; and
2. dampens the harmful effects of increased interpersonal conflict on weight by teaching participants how to induce a positive affect and self-affirming mindset

Participants in the control arm will receive the same number of lifestyle sessions as those randomized to the social network intervention.

Participants will:

1. Be randomly assigned to either the study group, which is asked to invite up to two friends or family members to join them at three coaching sessions, or the group that does not invite anyone.
2. Receive 15 coaching sessions over 24 weeks.
3. Complete an online questionnaire about eating and physical activity habits, confidence in developing healthier habits, mood, and health habits of twelve of their closest friends and family members.
4. Complete a 3-day weekly food log and wear a provided Fitbit for at least 9 hours daily.
5. The invited friends and family members will also be asked to complete a brief questionnaire about their eating and physical activity habits when they start and end the study.

ELIGIBILITY:
Inclusion Criteria:

* Index Participant:

  1. Black race or Hispanic ethnicity
  2. Male or Female 18 years of age or older
  3. Calculated BMI > 30kg/m2 from objectively measured height and weight by study staff
  4. Access & willingness to use program food intake app via home computer or a smartphone
  5. Ability to identify at least one adult social network member who will participate in the study
* Social Network Member:

  1. Male or Female 18 years of age or older
  2. Access to the internet or a smartphone

Exclusion Criteria:

* Index Participant:

  1. Active enrollment in a weight-loss program, use of weight-loss medications, or planning weight-loss surgery
  2. Advanced medical illness, dementia, hospitalization, injury, or pregnancy that inhibits regular physical activity
  3. Contraindications to exercise based on the Physical Activity Readiness Questionnaire or lack of clearance from a health care provider
  4. Unresolved Food insecurity
  5. Speaks a language other than English or Spanish
* Social Network Member:

  1. Speaks a language other than English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have attended at least 75 percent of the behavioral coaching sessions | End of study (24 weeks)
Number of intervention participants who have at least one social network member engage in the study | End of Study (24 weeks)
Number of participants and social network members combined who complete the final study assessment | End of Study (24 Weeks)

SECONDARY OUTCOMES:
Change in positive communication and problem solving as measured by the McMaster Family Assessment Device (FAD) Questionnaire | Baseline, End of Study (24 weeks)
  The lowest score on the McMaster Family Assessment Device (FAD) Questionnaire a participant can receive is 60 and the highest score on the McMaster Family Assessment Device (FAD) Questionnaire a participant can receive is 240. Higher scores mean positive family communication and problem solving.
Change in weight related social norms | Baseline, End of Study (24 weeks)
  A 5 point Likert scale that measures unhealthy weight norms. The lowest score is 7 and the highest score is 35. Higher scores mean healthy eating and physical activity weight norms.
Change in median Fitbit wear time in minutes | Weekly up to 24 weeks
  Total minutes spent in very active intensity during activity
Change in total caloric amounts on three-day food record | Weekly up to 24 weeks
  Participants complete food records at minimum 3 days a week
Change in median number of days that the Fitbit is worn | Weekly up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Erica G Phillips, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in any publication will be shared after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available beginning 6 months following publication and ending 5 years following publication.
Access Criteria: Anyone who wishes to access the data can request access for any purpose. Data will be made available and stored indefinitely in the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository.
URL: https://repository.niddk.nih.gov/pages/for_requestors/

REFERENCES:
- [Derived] Phillips E, Potter C, Poole J, Lewis A, Nahid M, Christos P, Hootman K, Winston G, de la Haye K. Reducing Obesity Using Social Ties (ROBUST): Protocol for a randomized control trial of a social network lifestyle intervention. PLoS One. 2025 Apr 16;20(4):e0318990. doi: 10.1371/journal.pone.0318990. eCollection 2025. PMID 40239159